CLINICAL TRIAL: NCT06309199
Title: Center of Excellence in Thai Pediatric Gastroenterology, Hepatology and Immunology
Brief Title: Prevalence of FGIDs and Probiotics Study
Acronym: PROOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Palittiya Sintusek, MD, Director, Head of Center of Excellence in Thai Pediatric Gastroenterology, Hepatology and Immunology, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0855/66
Record Dates: First submitted 2024-02-12; First posted 2024-03-13 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-08

CONDITIONS: Functional Gastrointestinal Disorders; Infant Conditions
Keywords: functional gastrointestinal disorder; colic; regurgitation; constipation; infant; prevalence
MeSH Terms: conditions — Gastrointestinal Diseases; Colic; Gastroesophageal Reflux; Constipation | interventions — Sunflower Oil

STUDY DESIGN:
Intervention Model Description: Intervention group received probiotics Control group received sunflower and MCT oil
Who Masked: Participant, Care Provider, Investigator
Masking Description: These 2 groups was assigned using computer generate with block of 4 and ratio 1:1.
  The intervention and placebo were prepare in the same container with the same color, odor and blinded to investigators, participants and guardians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics (Experimental): Limosilactobacillus reuteri DSM 17938 with sunflower oil and MCT oil were packed into a container. Infants will received 5 drops per day in the morning for 60 +/- 20 days
  Interventions: Dietary Supplement: Biogaia
- Placebo (Placebo Comparator): Sunflower oit and MCT oil were paced into a container. Infants will received 5 drops per day in the morning for 60+/- 20 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Biogaia — Biogaia is a probiotics product that contain Limosilactobacillus reuteri DSM 17938, sunflower oil and MCT oil
  Arms: Probiotics
Other: Placebo — Limosilactobacillus reuteri DSM 17938, sunflower oil and MCT oil
  Other Names: Sunflower oil + MCT oil
  Arms: Placebo

SUMMARY:
This is a study to evaluate the prevalence of FGIDs in infants using the Thai version of Rome IV diagnostic questionnaire for functional gastrointestinal disorders in infants and evaluate the efficacy of Limosilactobacillus reuteri DSM 17938 to prevent FGIDs in infants.

DETAILED DESCRIPTION:
This is a randomized controlled trial study about the the efficacy of Lactobacillus reuteri DSM 1987 to prevent FGIDs in healthy infants and the effect to gut microbiota diversity. The incidence of FGIDs in Thai infant using Thai version of ROME IV questionnaire (authorized by Rome Foundation) for infant and toddler and the associated factors of FGIDs also evaluate.

Population: target and control populations are the healthy infants born at King Chulalongkorn Memorial Hospital, Bangkok, Thailand, and can come to follow up at the hospital at 1, 2, 4, and 12 months of age Inclusion criteria

1. Healthy and term (GA 37-41 weeks) infants
2. Appropriate weight for age
3. APGAR score more than 8 at 10 minutes of life
4. Normal physical examination
5. Mothers have no previous probiotics use Methodology

   * Participants were double-blinded randomized using computer generation in block of four
   * Target population were received Limosilactobacillus reuteri DSM 17938 5 drops (0.185 mL) per day for 60 days
   * Control population were received mixture of sunflower oil and MCT oil 5 drop (0.185 mL) per day for 60 days
   * There were 5 visits at birth, 1, 2, 4, 12 months of life: the demographic data/Rome IV questionnaire for FGIDs in infant and associated factors with FGIDs record, physical examination and stool collection The study will be analyzed (open the randomized group) after all participants complete the 4-month follow-up period
   * Research assistance will telephone to them to take the Rome IV questionnaire for FGIDs at 3, 6, 9 months of life

Biological specimen collection Stool will be collected by rectal stimulation in each visit. The amount of >5 gm stool will be preserved in DNA and kept at -80 °C. All stool specimen will be processed the DNA extraction (DNA > 40 microlitre with concentration >50 ng/L). The DNA extraction for further amplification 16S rRNA using Illumina. The rest of the specimen will be kept up to 10 years for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy and term (GA 37-41 weeks) infants
2. Appropriate weight for age
3. APGAR score more than 8 at 10 minutes of life
4. Normal physical examination
5. Mothers have no previous probiotics use

Exclusion Criteria:

1. not willing to anticipate in the study
2. cannot come to follow-up until 1 year of age

Ages: 3 Days to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 512 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The prevalence of functional gastrointestinal disorders in the treatment group | at birth, 1 month, 2 months, 4 months
  Functional gastrointestinal disorders (colic, regurgitation, constipation, dyschazia and rumination) were assessed using the Thai version of Rome IV diagnostic questionnaire for neonates and toddlers

SECONDARY OUTCOMES:
The prevalence of functional gastrointestinal disorders in the placebo group | at birth, 1 month, 2 months, 4 months and 1 year (5-time points)
  Functional gastrointestinal disorders (include colic, regurgitation, constipation, dyschazia and rumination) were assessed using the Thai version of Rome IV diagnostic questionnaire for neonates and toddlers
The prevalence of functional gastrointestinal disorders in the treatment group | at 1 year of age
  Functional gastrointestinal disorders (colic, regurgitation, constipation, dyschazia and rumination) were assessed using the Thai version of Rome IV diagnostic questionnaire for neonates and toddlers

OTHER OUTCOMES:
Nutrition associated with functional gastrointestinal disorders in infants | at 1 year
  Amount of food composition (carbohydrate, protein, lipid - present as gm per kg body weight)
Gut microbial profiles associated with functional gastrointestinal disorder in infants | at birth, 1 month, 2 months, and 4 months
  Comparative metagenomic analysis of gut microbial profiles (diversity, relative abundance, species alteration) in fecal samples among different groups of infants
The sleep quality assessed by Brief Infant Sleep Revise Questionnaire of BISQR | at birth, 1 month, 2 months, 4 months and 1 year (5-time points)
  The questionnaire has 33 items in 3 main categories (Infant sleep, parent perception and parent behavior). Scores on each subscale and the total score are scaled from 0 to 100. Higher score denote better sleep quality.
Stool metabolomic substances (i.e microbial conjugation of secondary bile acid, aminoacid) and the stool metabolites alteration | at birth, 1 month, 2 months and 4 months
  Fecal metabolomic substances (i.e microbial conjugation of secondary bile acid, aminoacid) were assesse using liquid chromatography-mass spectrometry (LC-MS), gas chromatography-mass spectrometry (GC-MS) and capillary electrophoresis-mass spectrometry (CE-MS)
Fluid intake associated with functional gastrointestinal disorders in infants | at birth, 1 month, 2 months and 4 months and 1 year (5-time points)
  type of milk (breastfeeding or formula or mixed) and amount (mL per kg body weight)
Stress associated with functional gastrointestinal disorders in infants | at birth and 1 year
  stress in family (i.e divorce, family dept present as yes or no)
Antibiotics associated with functional gastrointestinal disorders in infants | at birth, 1 month, 2 months and 4 months and 1 year (5-time points)
  antibiotics use (yes or no)
Economic status associated with functional gastrointestinal disorders in infants | at birth and 1 year
  Economics status (income in baht)
Education of caregiver associated with functional gastrointestinal disorders in infants | at birth and 1 year
  Education (low, high)
Serious adverse effect during follow-up until end point | 1 month, 2 months, 4 months, 6 months, 9 months, 1 years
  admission, cause of admission, treatment details (intravenous fluid, medication, oxygen supplementation)
skin problems (seborrheic dermatitis, atopic dermatitis, nonspecific dermatitis) | 1 month, 2 months, 4 months, 1 year
  patient oriented- Scoring atopic dermatitis (it is an application in phone to add the information of skin lesion by doctor or parent examination), examination and record the characteristics and location of skin lesion by doctors

CONTACTS AND LOCATIONS:
Overall Officials: Yong Poovorawan, MD, Study Director — Center of Excellence in Clinical Virology
Locations (1):
- Maha Chakri Sirindhorn Clinical Research Center (Chula CRC), Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The data were collected anonymous.